CLINICAL TRIAL: NCT01740557
Title: A Pilot Study of Lymphodepletion Plus Adoptive Cell Transfer With T -Cells Transduced With CXCR2 and NGFR Followed by High Dose Interleukin-2 in Patients With Metastatic Melanoma
Brief Title: Genetically Modified Therapeutic Autologous Lymphocytes Followed by Aldesleukin in Treating Patients With Stage III or Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0471; NCI-2014-02655 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0471 (Other: M D Anderson Cancer Center); R01CA116206 (NIH)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (genetically modified T-cells, high-dose aldesleukin (Experimental): Patients receive cyclophosphamide IV over 2 hours on days -7 and -6, fludarabine phosphate IV daily over 15-30 minutes on days -5 to -1, and CXCR2-transduced autologous TIL and NGFR-transduced autologous TIL IV over up to 4 hours on day 0. Patients then receive high-dose aldesleukin IV over 15 minutes every 8-16 hours on days 1-5 (up to 15 doses) and 22-26 (up to 15 doses).
  Interventions: Biological: Aldesleukin; Biological: CXCR2-transduced Autologous Tumor Infiltrating Lymphocytes; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: NGFR-transduced Autologous T Lymphocytes; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: CXCR2-transduced Autologous Tumor Infiltrating Lymphocytes — Given IV
  Other Names: CXCR2-transduced Autologous TILs
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: NGFR-transduced Autologous T Lymphocytes — Given IV
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase I/II trial studies how well genetically modified therapeutic autologous lymphocytes (patient's own white blood cells) followed by aldesleukin work in treating patients with stage III melanoma or melanoma that has spread to other places in the body (metastatic). Placing chemokine (C-X-C motif) receptor 2 (CXCR2) and nerve growth factor receptor (NGFR) into lymphocytes (white blood cells) may help the body build an immune response to kill melanoma cells. Aldesleukin may enhance this effect by stimulating white blood cells to kill more melanoma cells. Giving genetically modified therapeutic autologous lymphocytes together with aldesleukin may be a better treatment for melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and safety of CXCR2 and NGFR transduced tumor-infiltrating lymphocytes (TIL) for treating metastatic malignant melanoma.

SECONDARY OBJECTIVES:

I. Determine whether CXCR2 transduction enhances the ability of TIL to migrate to melanoma tumors.

II. Determine the levels of CXCL1 and CXCL8 chemokines produced by melanoma tumors and assess whether this correlates with the tumor localization of CXCR2 transduced TIL.

III. Characterize the clinical response and correlate with migration of CXCR2 transduced TIL to the tumor and levels of CXCL1 and CXCL8 at the tumor site.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) over 2 hours on days -7 and -6, fludarabine phosphate IV daily over 15-30 minutes on days -5 to -1, and CXCR2-transduced autologous TIL and NGFR-transduced autologous TIL IV over up to 4 hours on day 0. Patients then receive high-dose aldesleukin IV over 15 minutes every 8-16 hours on days 1-5 (up to 15 doses) and 22-26 (up to 15 doses).

After completion of study treatment, patients are followed up at weeks 6 and 12, every 3 months for a year, and then annually for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* TURNSTILE I INCLUSION CRITERIA:
* Patients must have metastatic melanoma or stage III in-transit, subcutaneous, or regional nodal disease (Turnstile I)
* Patients must have a lesion amenable to resection for the generation of TIL (Turnstile I)
* Patients must receive a magnetic resonance imaging (MRI)/computed tomography (CT)/positron emission tomography (PET) of the brain within 6 months of signing informed consent; if new lesions are present, patient must have definitive treatment; principal investigator (PI) or his designee should make final determination regarding enrollment (Turnstile I)
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-2 within 30 days of signing informed consent (Turnstile I)
* Patients previously treated with immunotherapy, targeted therapy, or no therapy will be eligible; patients receiving cytotoxic agents will be evaluated by the PI or his designee
* Patients with a negative pregnancy test (urine or serum) must be documented within 14 days of screening for women of childbearing potential (WOCBP); a WOCBP has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months (Turnstile I)
* CHEMOTHERAPY/CELL INFUSION INCLUSION CRITERIA:
* Patients must have adequate TIL available (Turnstile II)
* Patients must have at least one biopsiable and measurable metastatic melanoma lesions >= 1 cm (Turnstile II)
* Patients may have brain lesions which measure =< 1 cm each (Turnstile II)
* Patients of both genders must practice birth control for four months after receiving the preparative regimen (lymphodepletion) and continue to practice birth control throughout the study; patients must have a documented negative pregnancy test (urine or serum) for women who have menstruation in the past 12 months and without sterilization surgery (Turnstile II)
* Unless surgically sterile by bilateral tubal ligation or vasectomy of partner(s), the patient agrees to continue to use a barrier method of contraception throughout the study such as: condom, diaphragm, hormonal, intrauterine device (IUD), or sponge plus spermicide; abstinence is an acceptable form of birth control (Turnstile II)
* Pregnancy testing will be performed within 14 days prior to treatment (Turnstile II)
* Clinical performance status of ECOG 0-2 within 14 days of lymphodepletion (Turnstile II)
* Absolute neutrophil count greater than or equal to 1000/mm^3 (Turnstile II)
* Platelet count greater than or equal to 100,000/mm^3 (Turnstile II)
* Hemoglobin greater than or equal to 8.0 g/dl (Turnstile II)
* Serum alanine transaminase (ALT) less than three times the upper limit of normal (Turnstile II)
* Serum creatinine less than or equal to 1.6 mg/dl (Turnstile II)
* Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's syndrome who must have a total bilirubin less than 3.0 mg/dl (Turnstile II)
* A stress cardiac test (stress thallium, stress multigated acquisition [MUGA] scan, dobutamine echocardiogram or other stress test that will rule out cardiac ischemia) within 6 months of lymphodepletion (Turnstile II)
* Forced expiratory volume in 1 second (FEV1) > 65% of predicted within 6 months of lymphodepletion (Turnstile II) or
* Forced vital capacity (FVC) > 65% of predicted within 6 months of lymphodepletion (Turnstile II)
* MRI/CT/PET of the brain within 30 days of lymphodepletion

Exclusion Criteria:

* Active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system; PI or his designee shall make the final determination regarding appropriateness of enrollment (Turnstile I)
* Patients who are pregnant or nursing (Turnstile I)
* CHEMOTHERAPY/CELL INFUSION EXCLUSION CRITERIA:
* Has had prior systemic cancer therapy within the past four weeks at the time of the start of the lymphodepletion regimen (Turnstile II)
* Women who are pregnant will be excluded (Turnstile II)
* Any active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, such as abnormal stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease; PI or his designee shall make the final determination regarding appropriateness of enrollment (Turnstile II)
* Any form of primary or secondary immunodeficiency; must have recovered immune competence after chemotherapy or radiation therapy as evidenced by lymphocyte counts (> 500/mm^3), white blood cell (WBC) (> 3,000/mm^3) or absence of opportunistic infections (Turnstile II)
* Requires no steroids within 4 weeks and have not used topical or inhalational steroids in the past 2 weeks prior to lymphodepletion; the exception being patients on chronic physiologic dose of steroid (Turnstile II)
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his designee, would prevent adequate informed consent or render immunotherapy unsafe or contraindicated (Turnstile II)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N Amaria, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Genetically Modified T-cells, High-dose Aldesleukin: Participants receive cyclophosphamide IV over 2 hours on days -7 and -6, fludarabine phosphate IV daily over 15-30 minutes on days -5 to -1, and CXCR2-transduced autologous TIL and NGFR-transduced autologous TIL IV over up to 4 hours on day 0. Participants then receive high-dose aldesleukin IV over 15 minutes every 8-16 hours on days 1-5 (up to 15 doses) and 22-26 (up to 15 doses).
  Aldesleukin: Given IV
  CXCR2-transduced Autologous Tumor Infiltrating Lymphocytes: Given IV
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  NGFR-transduced Autologous T Lymphocytes: Given IV
  Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Treatment (Genetically Modified T-cells, High-dose Aldesleukin
Started | 10
Completed | 8
Not Completed | 2
Not completed — Ineligible | 1
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Genetically Modified T-cells, High-dose Aldesleukin
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immune-Related Response
Description: Response will be defined as a 50% or greater decrease in the tumor's linear dimension post treatment, compared to baseline.
  Response will be evaluated by positron emission tomography or computed tomography imaging.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Genetically Modified T-cells, High-dose Aldesleukin
Number analyzed (Participants) | 8
Participants | 8

2. Primary Outcome: Number of Participants With Adverse Events Defined as Possible Grade 3 or Worse Toxicities
Description: Possible grade 3 or worse toxicities not normally associated with lymphodepletion and high dose IL-2 will be reported.
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Genetically Modified T-cells, High-dose Aldesleukin
Number analyzed (Participants) | 8
Participants | 8

3. Secondary Outcome: CXCR2 Transduction
Description: Determine whether CXCR2 transduction enhances the ability of TIL to migrate to melanoma tumors. his is a statistical version of the intuitive idea that, if the TIL methodology works as designed and the genetically transduced T-cells differentially recognize the cancer cell cytokines, then the ratio of post- and pre-treatment ratios RR = RY/RX should be larger than 1.
Time Frame: At infusion
Population: Data were not collected
Arm/Group | Treatment (Genetically Modified T-cells, High-dose Aldesleukin
Number analyzed (Participants) | 0

4. Secondary Outcome: CXCL1 and CXCL8 Chemokines Produced
Description: Determine the levels of CXCL1 and CXCL8 chemokines produced by melanoma tumors and assess whether this correlates with the tumor localization of CXCR2 transduced TIL
Time Frame: At infusion
Population: Data were not collected
Arm/Group | Treatment (Genetically Modified T-cells, High-dose Aldesleukin
Number analyzed (Participants) | 0

5. Secondary Outcome: Characterize the Clinical Response and Correlate With Migration of CXCR2 Transduced TIL to the Tumor and Levels of CXCL1 and CXCL8 at the Tumor Site.
Time Frame: At infusion
Population: Data were not collected
Arm/Group | Treatment (Genetically Modified T-cells, High-dose Aldesleukin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Baseline to 1 year follow-up
Arm/Group | Treatment (Genetically Modified T-cells, High-dose Aldesleukin
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Genetically Modified T-cells, High-dose Aldesleukin (N=8)
Death (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Fever (General disorders) | 4 (6)
Lung Infection (Infections and infestations) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Genetically Modified T-cells, High-dose Aldesleukin (N=8)
Abdominal Distension (Gastrointestinal disorders) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 7 (21)
Alanine aminotransferase increased (Investigations) | 2 (12)
Alkaline phosphatase increased (Investigations) | 5 (7)
Allergic Reaction (Immune system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9)
Anemia (Blood and lymphatic system disorders) | 7 (67)
Anorexia (Metabolism and nutrition disorders) | 7 (16)
Anxiety (Psychiatric disorders) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 6 (12)
Absolute monocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Absolute basophil cound decreased (Blood and lymphatic system disorders) | 1 (1)
Back Pain (right side lower back) (Musculoskeletal and connective tissue disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Bibasilar (Investigations) | 1 (1)
Blood bilirubin increased (Blood and lymphatic system disorders) | 8 (10)
Chills (General disorders) | 8 (20)
Constipation (Gastrointestinal disorders) | 5 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Creatinine increased (Investigations) | 5 (18)
Diarrhea (Gastrointestinal disorders) | 5 (9)
Diminished lung sounds- right (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Diminished lung sounds- left (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Diminished lung sound bilateral (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (6)
Dermititis (Skin and subcutaneous tissue disorders) | 2 (2)
Dark discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dysuria (Renal and urinary disorders) | 1 (1)
Edema Limbs (General disorders) | 4 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CK increased (Investigations) | 1 (1)
Decreased protein (Investigations) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Edema (face) (General disorders) | 1 (2)
Edema (trunk) (General disorders) | 1 (1)
ECG QT (Cardiac disorders) | 1 (1)
Elevated LDH (Investigations) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastitis (Gastrointestinal disorders) | 1 (1)
Tinea Cruris (fungal goin infection) (Infections and infestations) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Lung cracles- right (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythematous Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (Blood and lymphatic system disorders) | 7 (14)
Fever (General disorders) | 4 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (7)
Floaters (Gastrointestinal disorders) | 1 (1)
Generalised edema (Gastrointestinal disorders) | 1 (1)
Generalized erythema (General disorders) | 1 (1)
Generalized muscle weakness (General disorders) | 4 (6)
Headache (Nervous system disorders) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (16)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (16)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (11)
Hyponatremia (Metabolism and nutrition disorders) | 4 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (6)
Hypothyrodism (Endocrine disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INR Increased (Investigations) | 6 (11)
Insomnia (Psychiatric disorders) | 3 (3)
LDH Increased (General disorders) | 1 (4)
Lymphedema (Vascular disorders) | 2 (2)
Localized edema (Investigations) | 1 (1)
Ionized Calcium (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (17)
Ionized Calcium (Blood and lymphatic system disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Mucosal Infection (Gastrointestinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9)
Alkaline phosphate decreased (Blood and lymphatic system disorders) | 1 (7)
Oliguria (Investigations) | 1 (1)
Lung Infection (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Neutrophil count decreased (Investigations) | 8 (25)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 4 (5)
Palpitations (Cardiac disorders) | 1 (1)
Phosphorus increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 8 (54)
Platelet count increased (Investigations) | 1 (1)
Protein decreased (Investigations) | 1 (1)
Petechia (Skin and subcutaneous tissue disorders) | 2 (4)
Palpations (Cardiac disorders) | 1 (1)
Paresthesia (left shoulder) (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (bilateral hands/feet) (Nervous system disorders) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash masculo-papular (Skin and subcutaneous tissue disorders) | 3 (9)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (9)
Seizure (Nervous system disorders) | 1 (2)
Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Superventricular tachycardis (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Sommolence (Psychiatric disorders) | 1 (1)
Thrush (Gastrointestinal disorders) | 1 (1)
Total protein decreased (Metabolism and nutrition disorders) | 2 (3)
TSH increased (Investigations) | 2 (3)
Uric acid decreased (Blood and lymphatic system disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Weight gain (Investigations) | 4 (13)
Weight loss (Investigations) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
White blood cell decreased (Investigations) | 4 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT01740557/Prot_SAP_000.pdf